CLINICAL TRIAL: NCT05430464
Title: A Randomized, Controlled, Split Face Study of a 1726 nm Laser for the Treatment of Acne Vulgaris
Brief Title: A Study of a Laser for the Treatment of Acne Vulgaris
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cutera Inc. (Industry)
Collaborators: ethica Clinical Research Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: C-22-AC04
Record Dates: First submitted 2022-06-20; First posted 2022-06-24 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-09

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- 1726nm Laser Treatment (Experimental)
  Interventions: Device: 1726nm Laser System
- Sham Laser Treatment (Sham Comparator)
  Interventions: Device: Sham Laser System

INTERVENTIONS:
Device: 1726nm Laser System — Subjects will receive 1726nm laser treatments on one side of the face
  Arms: 1726nm Laser Treatment
Device: Sham Laser System — Subjects will receive sham laser treatments on the other side of the face.
  Arms: Sham Laser Treatment

SUMMARY:
The purpose of this study is to evaluate the onset, duration, efficacy and safety of the laser for the treatment of acne vulgaris.

ELIGIBILITY:
Inclusion Criteria:

* Female or Male, 16 to 50 years of age (inclusive).
* Fitzpatrick Skin Type I-VI
* Has clinically diagnosed acne vulgaris of moderate to severe on each hemiface and inflammatory acne lesions as determined by the blinded trained investigator (or qualified designee) using the Investigator's Global Assessment Scale.
* Subject (and legally authorized representative/substitute decision maker if subject is incapable of providing informed consent) must be able to read, speak, and understand English and sign the Informed Consent Form.
* Willing to stop using topical acne medications on the face for 2 weeks prior to baseline and systemic acne medications for 1 month prior to baseline and for the duration of the study.
* Willing and able to adhere to the treatment and follow-up schedule and pre/post-treatment care instructions.
* Willing to have very limited sun exposure (including avoiding tanning booths, sun lamps, sunbathing) and use an approved sunblock or sunscreen of SPF (Skin Protection Factor) 30 or higher on the face every day for the duration of the study, including the follow-up period.
* Willing to have photographs taken of the face and agree to the use of photographs for presentation, educational or marketing purposes.
* Agree to not undergo any other procedure(s) or add any new treatment modalities in the target area during the study.

Exclusion Criteria:

* Has clinically diagnosed acne vulgaris of severity grade of clear, almost clear, or mild on at least one hemiface as determined by the blinded trained investigator (or qualified designee) using the Investigator's Global Assessment Scale.
* Prior treatment to the target area during participation in a clinical trial of another device or drug within 1 month (30 days) prior to study participation.
* Prior treatment to the target area within 1 month of study participation including chemical peel, dermabrasion/microdermabrasion, microneedling, radiofrequency treatment, laser or light-based procedures, cryodestruction or chemodestruction, intralesional steroids, photodynamic therapy, or acne surgery.
* Prior injection of botulinum toxin in the target area within 1 month of study participation and for the duration of the study.
* Prior injection of collagen, hyaluronic acid filler or other dermal/tissue filler in the target area within 2 weeks of study participation.
* Systemic use of retinoid, such as isotretinoin, within 6 months of study participation.
* Started or changed hormonal contraception within 6 months of study participation or intends to start or change hormonal contraception through duration of the study. If subject has not changed hormonal contraception within 6 months of study participation and has intent of continuation through duration of this study, ok to enroll.
* History of malignant tumors in the target area.
* Excessive facial hair (e.g., beards, sideburns, moustaches, etc.) or facial adornments (studs, piercings, tattoos) that may preclude treatments, photos or accurate lesion assessments in the target area.
* Pregnant and/or breastfeeding or planning to become pregnant during the study.
* Presence of any skin condition in the target area (e.g., eczema, psoriasis, dermatitis, rash, papulo-pustular rosacea, infection) that would interfere with the diagnosis or assessment of acne vulgaris.
* Any medical condition that, in the opinion of the Investigator, would interfere with patient's participation in the full study protocol (e.g., severe Diabetes Mellitus or Cardiovascular Disease).
* Suffering from diagnosed coagulation disorders or taking prescription anticoagulation medications.
* History of diagnosed immunosuppression/immune deficiency disorders or currently using immunosuppressive medications.
* History of diagnosed connective tissue disease, such as systemic lupus erythematosus or scleroderma.
* Known hypersensitivity to, history of allergic reaction to, or contraindication to Pro-Nox (or similar) if administered.
* Any use of medication that is known to increase sensitivity to light according to Investigator's discretion.
* History of disease stimulated by heat, such as recurrent herpes simplex and/or herpes zoster (shingles) in the target area, unless treatment is conducted following a prophylactic regimen.
* History of radiation to the target area, currently undergoing treatment for skin cancer in the target area or undergoing systemic chemotherapy for the treatment of cancer.
* History of diagnosed pigmentary disorders (including vitiligo) in the target area.
* Facial tan or unable/unlikely to refrain from tanning on the face during the study.
* As per the Investigator's discretion, any physical or mental condition which might make it unsafe for the subject to participate in this study.

Ages: 16 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-07-27 (Actual); Primary Completion 2023-04 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Percent of subjects having at least a 1 point reduction on the Investigator Global Assessment Scale | 12 weeks

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Canadian Dermatology Centre, Toronto, Ontario
  - Windsor Clinical Research, Windsor, Ontario

IPD SHARING:
Plan to Share IPD: No